CLINICAL TRIAL: NCT06604117
Title: A Prospective, Open-label Study Evaluating the Effects of Probucol Combined with Statins on Atherosclerotic Characteristics and Prognosis in Patients with Ischemic Stroke
Brief Title: Efficacy of Probucol Combined with Statins Treatment for Ischemic Stroke
Acronym: EPCIS
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Xin Ma, Chief Doctor, Xuanwu Hospital, Beijing
Other Study IDs: IRB [2024]275-001
Record Dates: First submitted 2024-09-15; First posted 2024-09-19 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Ischemic Stroke; Atherosclerosis of Artery; Lipid Disorder; Statin
Keywords: Probucol; Statin; Atherosclerosis; Ischemic stroke; Plaque burden; Lipid-lowering treatment
MeSH Terms: conditions — Ischemic Stroke; Lipid Metabolism Disorders; Atherosclerosis | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Probucol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Conventional Lipid-Lowering Therapy Group: Participants who choose this group will receive conventional lipid-lowering therapy following current clinical guidelines, which may include statins, ezetimibe, or PCSK9 inhibitors. The treatment regimen will be tailored to the participants' individual needs but will not include Probucol.
  Interventions: Drug: Statin
- Combined Lipid-Lowering Therapy with Probucol Group: Participants who choose this group will receive a combination of conventional lipid-lowering therapy following current clinical guidelines (statins, ezetimibe, or PCSK9 inhibitors) and additional treatment with Probucol 0.5g twice daily. This regimen aims to further reduce atherosclerotic plaque burden and improve cardiovascular outcomes.
  Interventions: Drug: Probucol

INTERVENTIONS:
Drug: Statin — Participants who opt for this group will receive guideline-recommended conventional lipid-lowering therapy. For those with a history of ischemic stroke (IS), myocardial infarction (MI), acute coronary syndrome within the past year, symptomatic peripheral artery disease, or two or more high-risk factors, the target LDL-C level will be set at 1.4 mmol/L. For other IS participants, the LDL-C target will be set at 1.8 mmol/L. All participants will receive moderate-intensity statin therapy as the primary treatment. If LDL-C levels are not adequately controlled, ezetimibe will be added. If lipid levels remain unsatisfactory, the addition of PCSK9 inhibitors will be considered. Moderate-intensity statins are defined as atorvastatin 10-20 mg or rosuvastatin 5-10 mg.
  Other Names: Conventional Lipid-Lowering Therapy
  Groups: Conventional Lipid-Lowering Therapy Group
Drug: Probucol — Participants who choose this group will receive Probucol in combination with guideline-recommended lipid-lowering therapy. Specifically, participants in this group will take 0.5 grams of Probucol twice daily alongside the conventional lipid-lowering therapy mentioned in Group 1. The combination of Probucol and conventional therapy aims to further improve lipid profile and address atherosclerosis.
  Other Names: Probucol and Statin Combination Therapy
  Groups: Combined Lipid-Lowering Therapy with Probucol Group

SUMMARY:
The goal of this clinical trial is to evaluate whether the combination of Probucol with statin therapy can reduce the risk of vascular events and improve atherosclerosis outcomes in adults with ischemic stroke and confirmed atherosclerosis. The main questions it aims to answer are:

Does adding Probucol to statin therapy reduce plaque burden more effectively than statins alone? Does the combination therapy lead to fewer cardiovascular and cerebrovascular events compared to statins alone? Researchers will compare participants receiving standard statin therapy to those receiving statins combined with Probucol to assess differences in plaque burden and the occurrence of vascular events.

Participants will:

Choose either standard statin therapy (with possible addition of ezetimibe or PCSK9 inhibitors) or the same therapy combined with Probucol 0.5g twice daily.

Attend regular follow-up visits for monitoring atherosclerosis features and cardiovascular health over a 3-year period.

Undergo imaging studies to evaluate changes in atherosclerosis and blood tests to monitor lipid levels and other biomarkers.

DETAILED DESCRIPTION:
This single-center, prospective, open-label study will assess the effects of combining Probucol with statin therapy on the progression of atherosclerosis and the risk of vascular events in people with ischemic stroke. The primary hypothesis is that, in participants receiving guideline-recommended statin therapy, the addition of Probucol will reduce cardiovascular and cerebrovascular event risk, enhance plaque stability, and be well-tolerated.

The study will include participants aged 18 years or older who have experienced an ischemic stroke within the past 30 days and have confirmed atherosclerosis in any major artery (carotid, coronary, aortic, renal, or peripheral arteries). Participants will either follow a guideline-recommended lipid-lowering regimen (statins, with or without ezetimibe or PCSK9 inhibitors as needed) or a similar regimen combined with Probucol 0.5g twice daily. The study will enroll at least 100 participants in both the standard therapy group and the Probucol combination group.

Primary outcomes will include changes in plaque burden, while secondary outcomes will cover atherosclerotic features, composite vascular events (ischemic stroke, ischemic heart disease, vascular death), stroke recurrence, and poor functional prognosis (mRS ≥ 3). Exploratory outcomes will include changes in biochemical markers such as LDL-C, Ox-LDL, and Lp(a). Safety will be assessed by monitoring adverse events and serious adverse events.

Statistical analysis will include a multivariate linear regression model for primary outcomes, adjusted for baseline characteristics such as LDL-C levels and previous cardiovascular events. For time-to-event endpoints, Kaplan-Meier curves will be used, with Cox proportional hazards models providing hazard ratios. Subgroup analyses and repeated measures will further refine the understanding of treatment effects.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older.
2. Diagnosed with ischemic stroke (IS) confirmed by cranial CT/MRI.
3. Onset of stroke within the last 30 days.
4. Evidence of atherosclerosis (AS) in at least one artery (carotid, coronary, aorta, renal, or peripheral arteries) identified through neck CTA, coronary CTA, or ultrasound examination of lower extremity arteries.
5. Signed informed consent.

Exclusion Criteria:

1. History of allergy to Probucol or statins.
2. Non-atherosclerotic arterial stenosis, such as vasculitis, moyamoya disease, or arterial dissection.
3. Potential cardiac embolic sources, such as atrial fibrillation, artificial heart valves, endocarditis, or patent foramen ovale.
4. Known bleeding tendencies or hemorrhagic diseases, such as thrombocytopenia (platelet count < 100 × 10^9/L), hemorrhagic stroke, or gastrointestinal bleeding.
5. Severe myocardial diseases such as myocardial infarction (MI) or myocarditis.
6. Liver (ALT or AST > twice the upper limit of normal) or kidney (creatinine > 1.5 times the upper limit of normal or glomerular filtration rate < 50 ml/min) dysfunction.
7. Ventricular tachycardia, bradycardia, torsades de pointes, or syncopal episodes of cardiac origin.
8. Prolonged QT interval or conditions that may prolong the QT interval, such as certain medications.
9. Suffering from a severe illness with a life expectancy of less than one year or unable to cooperate due to cognitive or psychological issues.
10. Use of Probucol or any lipid-lowering medication other than statins, ezetimibe, and PCSK9 inhibitors within the 30 days prior to enrollment, including bile acid sequestrants, fibrates, and other similar drugs.
11. Pregnant or breastfeeding individuals, those trying to conceive.
12. Concurrent participation in another clinical trial involving investigational drugs or devices within the past 30 days.
13. Planned surgery or intervention that would require discontinuation of the study medication during the study period.
14. Any reason, known to the participant and investigator, that would prevent the participant from adhering to the study protocol or follow-up.
15. Other conditions determined by the investigator that may require exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of hospitalized individuals diagnosed with ischemic stroke at the Stroke Center of Xuanwu Hospital. Participants will be adults aged 18 years and older who meet the inclusion criteria specified for the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Change in Plaque Burden from Baseline to 12-Month Follow-up | Baseline to 12 months
  The primary outcome is the change in atherosclerotic plaque burden, measured as the percentage of stenosis at the most severe location of atherosclerotic plaque on computed tomography angiography (CTA). Plaque burden is calculated as 100% × (diameter of the plaque at its most severe point/diameter of the arterial lumen). The difference between the baseline and the 12-month follow-up measurement will be used to assess the effectiveness of the treatment.

SECONDARY OUTCOMES:
Change in High-Risk Plaque Count from Baseline to 12-Month Follow-up | Baseline to 12 months
  The change in the number of high-risk plaques in the coronary, aortic, and carotid arteries, assessed via CTA at the 12-month follow-up compared to baseline.
Change in Atherosclerotic Burden Score from Baseline to 12-Month Follow-up | Baseline to 12 months
  The change in the atherosclerotic burden score at 12 months, assessed through CTA imaging, compared to baseline. This score reflects the overall severity of atherosclerosis.
Occurrence of Cardiovascular Events at 12-Month and 24-Month Follow-up | 12 months and 24 months
  The incidence of composite cardiovascular events, including new fatal cardiovascular events, myocardial infarction (MI), unstable angina requiring hospitalization, and ischemic stroke (IS). Events will be reported based on whichever occurs first during the 12-month and 24-month follow-up.
Poor Functional Outcome at 1-Month Follow-up | 1 month and 3 months
  The occurrence of poor functional outcomes, defined as a modified Rankin Scale (mRS) score of ≥3, assessed during the first-month visit post-treatment.

OTHER OUTCOMES:
Changes in Biomarkers from Baseline to 12-Month Follow-up | Baseline to 12 months
  This outcome will assess the changes in various biochemical and inflammatory biomarkers from baseline to the 12-month follow-up. The biomarkers to be evaluated include:
  Low-Density Lipoprotein Cholesterol (LDL-C) High-Sensitivity C-Reactive Protein (hsCRP) Lipoprotein(a) [Lp(a)] Total Cholesterol Apolipoprotein B (ApoB) Apolipoprotein A1 (ApoA1) Other relevant biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Jing Dong, Doctor, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Xicheng District, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available from the corresponding author upon reasonable request after the publication of the study results. Data will not be shared prior to publication.

REFERENCES:
- [Background] Kong Q, Ma X, Wang C, Du X, Ren Y, Wan Y. Total Atherosclerosis Burden of Baroreceptor-Resident Arteries Independently Predicts Blood Pressure Dipping in Patients With Ischemic Stroke. Hypertension. 2020 Jun;75(6):1505-1512. doi: 10.1161/HYPERTENSIONAHA.120.15036. Epub 2020 Apr 27. PMID 32336234
- [Background] Arai H, Bujo H, Masuda D, Ishibashi T, Nakagawa S, Tanabe K, Kagimura T, Kang HJ, Kim MH, Sung J, Kim SH, Kim CH, Park JE, Ge J, Oh BH, Kita T, Saito Y, Fukushima M, Matsuzawa Y, Yamashita S. Integrated Analysis of Two Probucol Trials for the Secondary Prevention of Atherosclerotic Cardiovascular Events: PROSPECTIVE and IMPACT. J Atheroscler Thromb. 2022 Jun 1;29(6):850-865. doi: 10.5551/jat.62821. Epub 2021 Apr 18. PMID 33867420
- [Background] Li T, Chen W, An F, Tian H, Zhang J, Peng J, Zhang Y, Guo Y. Probucol attenuates inflammation and increases stability of vulnerable atherosclerotic plaques in rabbits. Tohoku J Exp Med. 2011 Sep;225(1):23-34. doi: 10.1620/tjem.225.23. PMID 21852751
- [Background] Naruszewicz M, Selinger E, Dufour R, Davignon J. Probucol protects lipoprotein (a) against oxidative modification. Metabolism. 1992 Nov;41(11):1225-8. doi: 10.1016/0026-0495(92)90013-z. PMID 1435295
- [Background] Zhu BB, Wang H, Chi YF, Wang YM, Yao XM, Liu S, Qiu H, Fang J, Yin PH, Zhang XM, Peng W. Protective effects of probucol on Ox-LDL-induced epithelial-mesenchymal transition in human renal proximal tubular epithelial cells via LOX-1/ROS/MAPK signaling. Mol Med Rep. 2018 Jan;17(1):1289-1296. doi: 10.3892/mmr.2017.7935. Epub 2017 Nov 2. PMID 29115480
- [Background] Mitra S, Deshmukh A, Sachdeva R, Lu J, Mehta JL. Oxidized low-density lipoprotein and atherosclerosis implications in antioxidant therapy. Am J Med Sci. 2011 Aug;342(2):135-42. doi: 10.1097/MAJ.0b013e318224a147. PMID 21747278
- [Background] Duarte Lau F, Giugliano RP. Lipoprotein(a) and its Significance in Cardiovascular Disease: A Review. JAMA Cardiol. 2022 Jul 1;7(7):760-769. doi: 10.1001/jamacardio.2022.0987. PMID 35583875
- [Background] Libby P. The changing landscape of atherosclerosis. Nature. 2021 Apr;592(7855):524-533. doi: 10.1038/s41586-021-03392-8. Epub 2021 Apr 21. PMID 33883728
- [Background] Kleindorfer DO, Towfighi A, Chaturvedi S, Cockroft KM, Gutierrez J, Lombardi-Hill D, Kamel H, Kernan WN, Kittner SJ, Leira EC, Lennon O, Meschia JF, Nguyen TN, Pollak PM, Santangeli P, Sharrief AZ, Smith SC Jr, Turan TN, Williams LS. 2021 Guideline for the Prevention of Stroke in Patients With Stroke and Transient Ischemic Attack: A Guideline From the American Heart Association/American Stroke Association. Stroke. 2021 Jul;52(7):e364-e467. doi: 10.1161/STR.0000000000000375. Epub 2021 May 24. No abstract available. PMID 34024117
- [Background] Khan SU, Yedlapati SH, Lone AN, Hao Q, Guyatt G, Delvaux N, Bekkering GET, Vandvik PO, Riaz IB, Li S, Aertgeerts B, Rodondi N. PCSK9 inhibitors and ezetimibe with or without statin therapy for cardiovascular risk reduction: a systematic review and network meta-analysis. BMJ. 2022 May 4;377:e069116. doi: 10.1136/bmj-2021-069116. PMID 35508321
- [Background] Libby P, Bornfeldt KE, Tall AR. Atherosclerosis: Successes, Surprises, and Future Challenges. Circ Res. 2016 Feb 19;118(4):531-4. doi: 10.1161/CIRCRESAHA.116.308334. No abstract available. PMID 26892955
- [Background] Virani SS, Newby LK, Arnold SV, Bittner V, Brewer LC, Demeter SH, Dixon DL, Fearon WF, Hess B, Johnson HM, Kazi DS, Kolte D, Kumbhani DJ, LoFaso J, Mahtta D, Mark DB, Minissian M, Navar AM, Patel AR, Piano MR, Rodriguez F, Talbot AW, Taqueti VR, Thomas RJ, van Diepen S, Wiggins B, Williams MS; Peer Review Committee Members. 2023 AHA/ACC/ACCP/ASPC/NLA/PCNA Guideline for the Management of Patients With Chronic Coronary Disease: A Report of the American Heart Association/American College of Cardiology Joint Committee on Clinical Practice Guidelines. Circulation. 2023 Aug 29;148(9):e9-e119. doi: 10.1161/CIR.0000000000001168. Epub 2023 Jul 20. PMID 37471501
- [Background] GBD 2019 Stroke Collaborators. Global, regional, and national burden of stroke and its risk factors, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Neurol. 2021 Oct;20(10):795-820. doi: 10.1016/S1474-4422(21)00252-0. Epub 2021 Sep 3. PMID 34487721
- [Background] Gutierrez J, Turan TN, Hoh BL, Chimowitz MI. Intracranial atherosclerotic stenosis: risk factors, diagnosis, and treatment. Lancet Neurol. 2022 Apr;21(4):355-368. doi: 10.1016/S1474-4422(21)00376-8. Epub 2022 Feb 7. PMID 35143758